CLINICAL TRIAL: NCT03247842
Title: The Analgesic and Rehabilitative Value of Supra-scapular Nerve Radiofrequency in Patients With Chronic Shoulder Pain After Breast Surgery.
Brief Title: The Analgesic Efficacy Supra-scapular Nerve RF After Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3024/01/15
Record Dates: First submitted 2017-04-24; First posted 2017-08-14 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain Syndrome
Keywords: post mastectomy pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprascapular nerve RF (Active Comparator): Eighty patients with chronic shoulder pain after breast surgery were allocated randomly into 2 groups (Figure1); forty patients received fluoroscopically guided supra-scapular nerve pulsed radiofrequency (PRF) followed by injection through the radiofrequency needle of mL of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group1)
  Interventions: Procedure: suprascapular nerve block
- suprascapular nerve block (Active Comparator): and forty patients received fluoroscopically guided supra-scapular nerve injection of mL of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group 2) without active pulsed radiofrequency only demo mode was applied.
  Interventions: Procedure: suprascapular nerve block

INTERVENTIONS:
Procedure: suprascapular nerve block — Sixty patients with shoulder dystocia after breast surgery will receive stellate ganglion neurolysis with supra-scapular nerve radiofrequency,

SUMMARY:
Eighty patients with chronic shoulder pain after breast surgery were allocated randomly into 2 groups; forty patients received fluoroscopically guided supra-scapular nerve pulsed radiofrequency (PRF) followed by injection of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group1) and forty patients received fluoroscopically guided supra-scapular nerve injection of of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group 2) without active pulsed radiofrequency only demo mode was applied.

DETAILED DESCRIPTION:
Eighty patients with chronic shoulder pain after breast surgery were allocated randomly into 2 groups ; forty patients received fluoroscopically guided supra-scapular nerve pulsed radiofrequency (PRF) followed by injection through the radiofrequency needle of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group1) and forty patients received fluoroscopically guided supra-scapular nerve injection of 0.25% bupivacaine solution containing 40 mg of methylprednisolone (group 2) without active pulsed radiofrequency only demo mode was applied.

ELIGIBILITY:
Inclusion Criteria:

* patients with post-mastectomy pain

Exclusion Criteria:

* Exclusion criteria are patients with any medical contraindications to neurolysis, patients with other bone metastases.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients with cancer breast
Enrollment: 80 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain | immedite postopertive
  assessment using visual analogue scale

SECONDARY OUTCOMES:
shoulder movement | 6 months after surgery
  shoulder mobility using long arm geniometry

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided